CLINICAL TRIAL: NCT03822897
Title: A Phase II Single Arm Trial of Elective Volume Adjusted De-Escalation Radiotherapy (EVADER) in Patients With Low-Risk HPV-Related Oropharyngeal Squamous Cell Carcinoma
Brief Title: De-Escalation Radiotherapy in Patients With Low-Risk HPV-Related Oropharyngeal Squamous Cell Carcinoma
Acronym: EVADER
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HN10
Record Dates: First submitted 2019-01-18; First posted 2019-01-30 (Actual); Results first posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Oropharyngeal Cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Radiation; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Other): This is a non-randomized, single-arm study evaluating elective volume-adjusted de-escalation radiotherapy. Patients receive one of two treatment options, based on treating physician discretion. Both options are considered part of a unified treatment strategy and analyzed as a single arm.
  * Option 1 (Chemoradiotherapy):
  Radiotherapy: 70 Gy to the high-risk volume and 56 Gy to the elective volume, delivered in 35 fractions over 7 weeks (5 fractions/week) Cisplatin: Either 100 mg/m² on days 1, 22, and 43 or 40 mg/m² weekly for 7 weeks
  * Option 2 (Radiotherapy Alone):
  Radiotherapy: 70 Gy to the high-risk volume and 56 Gy to the elective volume, delivered in 35 fractions over 6 weeks (6 fractions/week)
  Interventions: Radiation: Radiation; Drug: Cisplatin

INTERVENTIONS:
Radiation: Radiation — 35 fractions, 5/wk, 7 wks 70Gy/56Gy, or
  35 fractions, 6/wk, 6 wks, 70Gy/56Gy, or
  35 fractions, 5/wk, 7 wks OR 6/wk, 6 wks 70Gy/56Gy
  Other Names: No available
Drug: Cisplatin — 100 mg/m2 on day 1, 22, and 43 or 40 mg/m2 /wk for 7 wks
  Other Names: No available

SUMMARY:
The purpose of this study is to find out whether radiotherapy to some of the lymph node areas can be safely omitted to decrease side effects without increasing the risk of the tumour coming back.

DETAILED DESCRIPTION:
The standard or usual treatment for this disease includes radiotherapy or radiotherapy combined with chemotherapy or antibody therapy.

These treatments are highly effective at curing most patients with HPV-related cancer of the oropharynx, but short and long-term side effects from treatment can be significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically proven diagnosis of HPV-related OPSCC
* Clinical stage T1-3 N0-1 M0 (UICC/AJCC 8th Ed.)
* Patients must be eligible for definitive RT or CRT
* Must be ≥ 18 years of age
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Patient is able (i.e. sufficiently fluent) and willing to complete the quality of life and health economics questionnaires in either English or French
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrolment in the trial to document their willingness to participate
* Patients must be accessible for treatment and follow-up. Investigators must assure themselves the patients enrolled on this trial will be available for complete documentation of the treatment, adverse events, and follow-up.
* In accordance with CCTG policy, protocol treatment is to begin within 3 weeks of patient registration
* Women/men of childbearing potential must have agreed to use a highly effective contraceptive method
* The following radiological investigations must be done within 8 weeks of randomization: CT or MR of head and neck (MRI is recommended for base-of-tongue primary tumors); PET-CT scan.
* Patient must consent to provision of, and investigator(s) must confirm location and commit to obtain a representation of formalin-fixed paraffin block of non-cytology tumour tissue in order that the specific correlative marker assays described in Section 12 (Correlative Studies) may be conducted. Please see the Correlative Manual for details
* Patient must consent to provision of samples of blood and plasma (for circulating cell free DNA) in order that the specific correlative marker assays described may be conducted.
* Patients with prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.

Exclusion Criteria:

* Previous chemotherapy or radiotherapy treatment for head and neck cancer
* Patients with an unknown primary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Bratman, Study Chair — Princess Margaret Cancer Centre, Toronto, ON
Locations (14):
- Canada (14):
  - BCCA - Centre for the North, Prince George, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - The Jewish General Hospital, Montreal, Quebec
  - The Research Institute of the McGill University, Montreal, Quebec
  - Hotel-Dieu de Quebec, Québec, Quebec
  - CIUSSS de l'Estrie - Centre hospitalier, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Arm: Elective volume adjusted de-escalation radiotherapy.
  Option #1 - Radiotherapy 35 fractions, 5/wk, 7 wks 70Gy/56Gy Cisplatin 100mg/m2 on day 1, 22 and 43 or 40mg mg/m2/wk for 7 wks
  Option #2 - Radiation only-35 fraction, 6/wk, 6wks 70Gy/56Gy
Period: Overall Study
Arm/Group | Experimental Arm
Started | 103
Completed | 100
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Experimental Arm
Number analyzed (Participants) | 103
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62.8 [56 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 85
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
ECOG Performance Status [Count of Participants; unit: Participants] — The ECOG Performance Status is a scale used to assess a patient's level of functioning. ECOG 0 indicates the patient fully active, able to carry on all pre-disease performance without restriction; ECOG 1 means the patient is restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g. light housework, office work.
  Participants
    0 | 82
    1 | 21

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival
Description: Event free survival (EFS) is defined as the time from the date of registration to the date of first record of any of the following events:
  * Progression.
  * Surgery.
  * Non-protocol RT, chemotherapy, or biologic therapy (for the current cancer diagnosis) without documentation of the site of failure.
  * Death due to any cause. The outcome is reported as the proportion of patients who remain event-free at 2 years.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: Percentage of patients event-free at 2y
Arm/Group | Experimental Arm
Number analyzed (Participants) | 99
Percentage of patients event-free at 2y | 91.8 [86.6 to 97.4]

2. Secondary Outcome: Overall Survival
Description: For patients who have died, overall survival is calculated in months from the day of registration to date of death. Otherwise, overall survival is censored at the last day the patient is known alive (LKA). The outcome is reported as the proportion of patients who remain alive at 2 years.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: Percentage of patients alive at 2 years
Arm/Group | Experimental Arm
Number analyzed (Participants) | 99
Percentage of patients alive at 2 years | 94.7 [90.2 to 99.3]

3. Secondary Outcome: Local-regional Control
Description: Local-regional control is defined as the time from the date of registration to the date of any of the following, whichever comes first:
  * Surgery of primary tumour at any time performed for clinical or radiological disease persistence/progression/recurrence with tumour present/unknown on final pathology.
  * Neck dissection > 20 weeks from the end of radiation therapy performed for clinical or radiological (RECIST 1.1) disease persistence/progression/recurrence within target volumes with tumour present/unknown on final pathology.
  * Neck dissection at any time after registration performed for clinical or radiological disease recurrence/progression outside the target volumes or without documentation of the site of failure with tumour present/unknown on final pathology.
  * the first record of appearance (radiological or clinical) of local or regional disease progression. The outcome is reported as the proportion of patients who remain local-regional control free at 2 years.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: Percentage of patients LRC free at 2y
Arm/Group | Experimental Arm
Number analyzed (Participants) | 99
Percentage of patients LRC free at 2y | 94.8 [90.5 to 99.3]

4. Secondary Outcome: Out-of-field Regional Control
Description: Time to out-of-field regional failure is defined as the time from the date of registration to the date of the first record of appearance of regional progression/recurrence outside the treatment field , or to the date of neck dissection at any time after registration with tumour present/unknown performed for clinical or radiological disease progression outside the target volumes whichever comes first. The outcome is reported as the proportion of patients who remain out-of-field regional control free at 2 years.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: Percentages of patients ORC free at 2y
Arm/Group | Experimental Arm
Number analyzed (Participants) | 99
Percentages of patients ORC free at 2y | 99 [97 to 100]

5. Secondary Outcome: Distant Metastasis Free Survival
Description: Distant metastasis free survival is defined as the time from the date of registration to the date of first record of appearance of distant metastasis or death for any cause. Local-regional failure or second cancers diagnosed before the distant metastases are not considered events of interest for this endpoint. Subjects alive and free of distant metastasis are censored at the date of the most recent follow-up examination. The outcome is reported as the proportion of patients who remain distant metastasis event-free at 2 years.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: Percentages of patients DMF at 2y
Arm/Group | Experimental Arm
Number analyzed (Participants) | 99
Percentages of patients DMF at 2y | 91.3 [84.7 to 98.3]

ADVERSE EVENTS:
Time Frame: Adverse events are assessed weekly during protocol therapy, then at 1, 3, 6, 9, 12, 15, 18, 21, 24, 28, 32, and 36 months post-radiotherapy, then every 6 months until 60 months post-radiotherapy or until recurrence/progression, and as clinically indicated thereafter.
Description: Adverse events were collected and reported for all patients as a single group, without distinction between the two radiotherapy delivery options.
Arm/Group | Experimental Arm
All-Cause Mortality (participants affected / at risk) | 6/100
Serious Adverse Events (participants affected / at risk) | 8/100
Other Adverse Events (participants affected / at risk) | 100/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Arm (N=100)
Dysphagia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Other gastrointestinal disorders (Gastrointestinal disorders) | 1
Lung infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Acute kidney injury (Renal and urinary disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Arm (N=100)
Ear pain (Ear and labyrinth disorders) | 14
Hearing impaired (Ear and labyrinth disorders) | 6
Tinnitus (Ear and labyrinth disorders) | 26
Constipation (Gastrointestinal disorders) | 39
Diarrhea (Gastrointestinal disorders) | 6
Dry mouth (Gastrointestinal disorders) | 94
Dysphagia (Gastrointestinal disorders) | 49
Mucositis oral (Gastrointestinal disorders) | 82
Nausea (Gastrointestinal disorders) | 36
Oral pain (Gastrointestinal disorders) | 23
Salivary duct inflammation (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 16
Other gastrointestinal disorders (Gastrointestinal disorders) | 34
Fatigue (General disorders) | 52
Neck edema (General disorders) | 6
Pain (General disorders) | 9
Thrush (Infections and infestations) | 10
Dermatitis radiation (Injury, poisoning and procedural complications) | 78
Neutrophil count decreased (Investigations) | 8
Weight loss (Investigations) | 34
Anorexia (Metabolism and nutrition disorders) | 24
Dehydration (Metabolism and nutrition disorders) | 13
Neck pain (Musculoskeletal and connective tissue disorders) | 12
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 19
Dizziness (Nervous system disorders) | 11
Dysgeusia (Nervous system disorders) | 86
Headache (Nervous system disorders) | 8
Paresthesia (Nervous system disorders) | 9
Peripheral sensory neuropathy (Nervous system disorders) | 6
Anxiety (Psychiatric disorders) | 13
Insomnia (Psychiatric disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Hiccups (Respiratory, thoracic and mediastinal disorders) | 6
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 12
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 17
Sore throat (Respiratory, thoracic and mediastinal disorders) | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/97/NCT03822897/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-16): https://cdn.clinicaltrials.gov/large-docs/97/NCT03822897/SAP_001.pdf